CLINICAL TRIAL: NCT04634682
Title: Assessing the Effect of the MYODM Food Supplement on Quality of Life, Fatigue and Hypersomnia in Patients With Myotonic Dystrophy Type 1
Brief Title: Effect of MYODM on Quality of Life, Fatigue and Hypersomnia in Patients With Myotonic Dystrophy Type 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Myogem Health Company, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RFT-MYO-2020-01
Record Dates: First submitted 2020-09-25; First posted 2020-11-18 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Myotonic Dystrophy 1
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MYODM (Experimental): MYODM, three times a day, orally
  Interventions: Dietary Supplement: MYODM
- No intervention (No Intervention): Patients will follow the same evaluation schedule but will not receive MYODM

INTERVENTIONS:
Dietary Supplement: MYODM — Formulated composition containing Theobroma cacao supplemented with caffeine
  Arms: MYODM

SUMMARY:
The purpose of this study is to determine whether MYODM (formulated composition containing Theobroma cacao supplemented with caffeine (caffeine/theobromine ratio1/1.85, w/w) is effective in the treatment of excessive daytime sleepiness due to myotonic dystrophy type 1 (DM1) and improves the quality of life of these patients.

DETAILED DESCRIPTION:
Detailed Description:

Myotonic Dystrophy type I (DM1) is the most common form of adult muscular dystrophy, affecting 1 in 8000 individuals. It is an autosomal dominant disorder with multisystemic involvement of multiple organs and tissues, mainly brain, heart, endocrine system, eyes and both smooth and skeletal muscles.

Hypersomnolence is one of the most frequently reported symptoms in patients with DM1 and often lead to handicap such as cessation of employment and withdrawal from social activities. The present project is a 6 month randomized study to assess the effect of MYODM on fatigue, hypersomnia and quality of life in DM1 patients.The patients will be randomized to one of the two study arms. The active arm will receive the MYODM treatment and the control arm will not but both will follow the same evaluation program.

Patients will come to the center every 3 months for evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Genetically proven DM1
* Able to walk independently

Exclusion Criteria:

* Regular intake of plant stanols or other nutritional supplement
* Co-morbidity interfering with the interventions or possibly influencing outcomes.
* Participation in another clinical trial at the same time
* Unable to complete study questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Change in Individualized Neuromuscular Quality of Life (INQoL) Mean Scores | Screening, Month 3, Month 6
  Scores from the self-administered INQoL questionnaire will be compared at the start of the study (Month 0) and at the end (Month 6) among the MYODM treated group and the control group. Scores range from 0-100, with 100 being a better outcome.
Change in Individualized Short Form-36 (SF-36) Mean Scores | Screening, Month 3, Month 6
  Scores from the self-administered SF-36 questionnaire will be measured at the start of the study (Month 0), and at the end (Month 6) among patients in the MYODM-treated group and control group. Mean scores range from 0 (minimum) - 100 (maximum) with higher mean scores reflecting better outcomes.
Change in Epworth Sleepiness Scale (ESS) Scores | Screening, Month 3, Month 6
  ESS score range is 0-24; lower ESS scores indicate less daytime sleepiness; higher ESS scores indicate more severe sleepiness

SECONDARY OUTCOMES:
Change in Physical activity and daytime sleepiness measured with GeneActiv actometer | Screening, Baseline, Month 6

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Donostia, San Sebastián, Guipuzkoa, Spain